CLINICAL TRIAL: NCT01593566
Title: Femoral Nerve Block Using 0.25% Versus 0.5% Bupivacaine for Analgesia After Arthroscopic Anterior Cruciate Ligament Reconstruction
Brief Title: Femoral Nerve Block for Analgesia After Anterior Cruciate Ligament Reconstruction
Acronym: FNB for ACLR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, arissara iamaroon, associated professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mahidol University
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Analgesia After ACL Reconstruction
Keywords: femoral nerve block
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.25% bupivacaine (Active Comparator): femoral nerve block using 0.25% bupivacaine versus 0.5% bupivacaine
  Interventions: Drug: 0.25% Bupivacaine
- 0.5% bupivacaine (Active Comparator): femoral nerve block using 0.25% bupivacaine versus 0.5% bupivacaine
  Interventions: Drug: 0.5% Bupivacaine

INTERVENTIONS:
Drug: 0.25% Bupivacaine — Femoral nerve block using 0.25% versus 0.5% bupivacaine
  Other Names: marcaine
  Arms: 0.25% bupivacaine
Drug: 0.5% Bupivacaine — Femoral nerve block using 0.25% versus 0.5% bupivacaine for analgesia after ACL reconstruction
  Other Names: marcaine
  Arms: 0.5% bupivacaine

SUMMARY:
Femoral nerve block using 0.25% bupivacaine or 0.5% bupivacaine provides a longer time for analgesia after Anterior Cruciate Ligament (ACL) reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for ACL reconstruction
* ASA physical status I-II
* Body weight > or = 50 kg.

Exclusion Criteria:

* Patients with redo ACL reconstruction
* Contraindication to neuraxial block
* allergy to local anesthetics, sulfa, NSAIDs, morphine, paracetamol
* Patients with communication problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
time to first analgesic requirement | 48 hr

SECONDARY OUTCOMES:
pain score scale | 48 hr

CONTACTS AND LOCATIONS:
Overall Officials: arissara iamaroon, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand